CLINICAL TRIAL: NCT04178096
Title: Using Data-Driven Implementation Strategies to Improve the Quality of Cirrhosis Care (PEC 19-307)
Brief Title: Using Data-Driven Implementation Strategies to Improve the Quality of Cirrhosis Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: VA Pittsburgh Healthcare System (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: PEX 19-003; 1I50HX002903-01A1 (NIH)
Record Dates: First submitted 2019-11-06; First posted 2019-11-26 (Actual); Results first posted 2025-04-01 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: Cirrhosis, Liver
Keywords: Hepatitis C; Liver Diseases; Hepatitis; Virus Diseases; Cirrhosis, Liver; Liver Cirrhoses; Hepatic Cirrhoses; Implementation Science; Strategies; Evaluation
MeSH Terms: conditions — Liver Cirrhosis; Hepatitis C; Liver Diseases; Hepatitis; Virus Diseases

STUDY DESIGN:
Intervention Model Description: The investigators will select 'low-performing' sites to receive a bundle of strategies that have been empirically determined to be associated with evidence based practices for Veterans with cirrhosis. Using a hybrid type III stepped wedge cluster design, in which the investigators provide the bundle of strategies to four sites every six month period, then will evaluate whether applying these data-driven implementation strategies increases the use of evidence based practices and outcomes for cirrhosis compared to VA sites operating as usual.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Quality Improvement Intervention (Other): Low-performing sites will receive a package of strategies which have been empirically determined to be associated with successful implementation of evidence based practices that lead to improved health outcomes for Veterans with cirrhosis. This stepped wedge trial cluster randomized patients to the timing of site-level intervention.
  Interventions: Other: Quality Improvement Intervention

INTERVENTIONS:
Other: Quality Improvement Intervention — The investigators will assess the effectiveness of empirically determined implementation strategies that are associated with increasing cirrhosis evidence based practices and thus improving outcomes of Veterans with cirrhosis by introducing a bundle of these strategies to four new 'low-performing' hospitals every six months during and eighteen month period in this stepped wedge cluster randomized trial.

SUMMARY:
This Veteran Affairs (VA) Quality Improvement project aims to understand which data-driven implementation strategies promote evidence based practices that improve high-quality care for Veterans with cirrhosis.

DETAILED DESCRIPTION:
Nearly 120,000 Veterans in care have cirrhosis, or advanced liver disease, from alcohol, hepatitis C, fatty liver disease, or other causes, and this number is rapidly increasing. There are life-saving measures that providers can take to prevent harm from cirrhosis. The three most impactful of these measures include providing access to post-discharge follow-up and screening for liver cancer and esophageal varices (veins that can cause catastrophic bleeding). However, only about one-third of Veterans receive care aligned with these three evidence-based practices (EBPs). Therefore, there is an urgent need to improve access to high-quality care for Veterans with this common condition.

By focusing on strategies that most successfully encourage implementation of evidence-based practices the investigators can address the urgent need to improve the quality and timeliness of care for Veterans with cirrhosis who receive care at VA hospitals. This quality improvement intervention seeks to understand which implementation strategies, or discrete activities that are conducted to promote EBP implementation, improve cirrhosis care. The aims of this evaluation are to: (1) empirically determine which combinations of implementation strategies ('data-driven strategies') are associated with the successful implementation of EBPs for Veterans with cirrhosis, (2) use Intervention Mapping to operationalize the 'data-driven' implementation strategies developed in the first aim, and (3) evaluate whether applying data-driven implementation strategies increases the use of EBPs for cirrhosis, using a hybrid type III stepped wedge cluster randomized trial. The investigators will measure cirrhosis care at all VA sites and use the data from aims 1 and 2 to provide feedback to all sites. The investigators anticipate that more intensive implementation interventions will directly impact 12 of the lowest-performing sites.

ELIGIBILITY:
Inclusion Criteria:

* Veterans who have cirrhosis, or advanced liver disease, and receive care at VA.

Exclusion Criteria:

* N/A

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2020-09-18 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shari S Rogal, MD MPH, Principal Investigator — VA Pittsburgh Healthcare System University Drive Division, Pittsburgh, PA
Locations (1):
- VA Pittsburgh Healthcare System University Drive Division, Pittsburgh, PA, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Yakovchenko V, Kang C, Neely B, Lamorte C, McCurdy H, Scott D, Nobbe A, Robins G, Ekanem NR, Merante M, Gibson S, Spoutz P, Chia L, Gonzalez RI, Chinman MJ, Ross D, Chartier M, Beste LA, Bajaj JS, Taddei T, Morgan TR, Rogal SS. Getting to Implementation: applying data-driven implementation strategies to improve guideline concordant surveillance for hepatocellular carcinoma. Implement Sci. 2025 Dec 12;20(1):53. doi: 10.1186/s13012-025-01469-w. PMID 41388318
- [Derived] Yakovchenko V, Merante M, Chinman MJ, Neely B, Lamorte C, Gibson S, Kirchner J, Morgan TR, Rogal SS. The "good enough" facilitator: elucidating the role of working alliance in the mechanism of facilitation. Implement Sci Commun. 2025 Feb 25;6(1):22. doi: 10.1186/s43058-025-00705-0. PMID 40001234
- [Derived] Yakovchenko V, Rogal SS, Goodrich DE, Lamorte C, Neely B, Merante M, Gibson S, Scott D, McCurdy H, Nobbe A, Morgan TR, Chinman MJ. Getting to implementation: Adaptation of an implementation playbook. Front Public Health. 2023 Jan 6;10:980958. doi: 10.3389/fpubh.2022.980958. eCollection 2022. PMID 36684876
- [Derived] Rogal SS, Yakovchenko V, Morgan T, Bajaj JS, Gonzalez R, Park A, Beste L, Miech EJ, Lamorte C, Neely B, Gibson S, Malone PS, Chartier M, Taddei T, Garcia-Tsao G, Powell BJ, Dominitz JA, Ross D, Chinman MJ. Getting to implementation: a protocol for a Hybrid III stepped wedge cluster randomized evaluation of using data-driven implementation strategies to improve cirrhosis care for Veterans. Implement Sci. 2020 Oct 21;15(1):92. doi: 10.1186/s13012-020-01050-7. PMID 33087156

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: sites
Groups:
- Round 1 (Oct 2020-Mar 2021); Round 2 (Apr 2021-Sep 2021); Round 3 (Oct 2021-Mar 2022): Low-performing sites will receive a package of strategies which have been empirically determined to be associated with successful implementation of evidence based practices that lead to improved health outcomes for Veterans with cirrhosis.
  Quality Improvement Intervention: The investigators will assess the effectiveness of empirically determined implementation strategies that are associated with increasing cirrhosis evidence based practices and thus improving outcomes of Veterans with cirrhosis by introducing a bundle of these strategies to four new 'low-performing' hospitals every six months during an eighteen month period in this stepped wedge cluster randomized trial.
Period: Oct 2020-Mar 2021
Arm/Group | Round 1 (Oct 2020-Mar 2021) | Round 2 (Apr 2021-Sep 2021) | Round 3 (Oct 2021-Mar 2022)
Started | NA; 4 sites (Individual participants were not enrolled.) | NA; 0 sites (Individual participants were not enrolled.) | NA; 0 sites (Individual participants were not enrolled.)
Completed | NA; 4 sites (Individual participants were not enrolled.) | NA; 0 sites (Individual participants were not enrolled.) | NA; 0 sites (Individual participants were not enrolled.)
Not Completed | NA; 0 sites | NA; 0 sites | NA; 0 sites
Period: Apr 2021-Sep 2021
Arm/Group | Round 1 (Oct 2020-Mar 2021) | Round 2 (Apr 2021-Sep 2021) | Round 3 (Oct 2021-Mar 2022)
Started | NA; 0 sites (Individual participants were not enrolled.) | NA; 4 sites (Individual participants were not enrolled.) | NA; 0 sites (Individual participants were not enrolled.)
Completed | NA; 0 sites (Individual participants were not enrolled.) | NA; 3 sites (Individual participants were not enrolled.) | NA; 0 sites (Individual participants were not enrolled.)
Not Completed | NA; 0 sites | NA; 1 sites | NA; 0 sites
Period: Oct 2021-Mar 2022
Arm/Group | Round 1 (Oct 2020-Mar 2021) | Round 2 (Apr 2021-Sep 2021) | Round 3 (Oct 2021-Mar 2022)
Started | NA; 0 sites (Individual participants were not enrolled.) | NA; 0 sites (Individual participants were not enrolled.) | NA; 4 sites (Individual participants were not enrolled.)
Completed | NA; 0 sites (Individual participants were not enrolled.) | NA; 0 sites (Individual participants were not enrolled.) | NA; 3 sites (Individual participants were not enrolled.)
Not Completed | NA; 0 sites | NA; 0 sites | NA; 1 sites

BASELINE CHARACTERISTICS:
Population: Individual participants were not enrolled.
Groups:
- Quality Improvement Intervention: Low-performing sites will receive a package of strategies which have been empirically determined to be associated with successful implementation of evidence based practices that lead to improved health outcomes for Veterans with cirrhosis.
  Quality Improvement Intervention: The investigators will assess the effectiveness of empirically determined implementation strategies that are associated with increasing cirrhosis evidence based practices and thus improving outcomes of Veterans with cirrhosis by introducing a bundle of these strategies to four new 'low-performing' hospitals every six months during and eighteen month period in this stepped wedge cluster randomized trial.
Arm/Group | Quality Improvement Intervention
Number analyzed (Participants) | 0
Age, Categorical
Age, Continuous
Sex: Female, Male
Race (NIH/OMB)
Region of Enrollment [unit: participants]

OUTCOME MEASURES:

1. Primary Outcome: Hepatocellular Carcinoma Screening
Description: Active patients, or those with outpatient or prescription activity within the last eighteen months, with a diagnosis of cirrhosis should have abdominal imaging every 6 months. Hepatocellular carcinoma (HCC) and Post-transplant patients are not included. This measure is being assessed by comparing the patients that have had imaging for liver cancer screening in the last eight months to those that have not.
Time Frame: 6 months after the previous screening.
Measure: Number (95% Confidence Interval); unit: Odds ratio
Arm/Group | Quality Improvement Intervention
Number analyzed (Participants) | 8243
Odds ratio | 1.61 [1.54 to 1.69]

ADVERSE EVENTS:
Time Frame: 1 year
Description: Individual participants were not enrolled. "Participants" here refers to sites.
Arm/Group | Quality Improvement Intervention
All-Cause Mortality (participants affected / at risk) | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12
Other Adverse Events (participants affected / at risk) | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2021-09-09): https://cdn.clinicaltrials.gov/large-docs/96/NCT04178096/Prot_000.pdf
  • Statistical Analysis Plan (2024-12-30): https://cdn.clinicaltrials.gov/large-docs/96/NCT04178096/SAP_001.pdf